CLINICAL TRIAL: NCT01354353
Title: Safety and Tolerability of Multiple Ascending Doses of LY2140023 in Subjects With Schizophrenia
Brief Title: A Study of Safety and Tolerability in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13565; H8Y-MC-HBDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; pomaglumetad methionil; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Aripiprazole (Active Comparator): Part A: Continue current prescribed dosing regimen -- Study Day 1 to discharge (Study Day 21). Part B: Continue current prescribed dosing regimen (≤ 30 milligrams [mg]/day ) -- Study Day 1 to discharge (Study Day 23, 25 or 28 based on adaptive design)
  Interventions: Drug: Aripiprazole
- Part A: 160 mg LY2140023 (Experimental): Administered orally, twice daily (BID) for 6 days (Study Days 10-15) and as a single morning dose on the 7th day (Study Day 16)
  Interventions: Drug: LY2140023
- Part A: 240 mg LY2140023 (Experimental): Administered orally BID for 6 days (Study Days 10-15) and as a single morning dose on the 7th day (Study Day 16)
  Interventions: Drug: LY2140023
- Part A: 320 mg LY2140023 (Experimental): Administered orally BID for 6 days (Study Days 10-15) and as a single morning dose on the 7th day (Study Day 16)
  Interventions: Drug: LY2140023
- Part A: 400 mg LY2140023 (Experimental): Administered orally BID for 6 days (Study Days 10-15) and as a single morning dose on the 7th day (Study Day 16)
  Interventions: Drug: LY2140023
- Part A: 480 mg LY2140023 (Experimental): Administered orally BID for 6 days (Study Days 10-15) and as a single morning dose on the 7th day (Study Day 16)
  Interventions: Drug: LY2140023
- Part B: LY2140023 (Experimental): If doses up to or equal to 400 mg BID are not tolerated, Part B of the study may be started. The dose of LY2140023 will be titrated in the same participant from highest dose that was tolerated in Part A, with the intention to reach a dose of 480 mg LY2140023.
  Interventions: Drug: LY2140023

INTERVENTIONS:
Drug: LY2140023 — Administered orally
  Other Names: pomaglumetad methionil
  Arms: Part A: 160 mg LY2140023; Part A: 240 mg LY2140023; Part A: 320 mg LY2140023; Part A: 400 mg LY2140023; Part A: 480 mg LY2140023; Part B: LY2140023
Drug: Aripiprazole — Administered orally
  Other Names: Abilify
  Arms: Aripiprazole

SUMMARY:
This is an inpatient, open-label, multiple-dose, multicenter study to evaluate the safety and tolerability of LY2140023 given at doses expected to reflect multiples of the anticipated therapeutic exposure under clinical investigation. In the event of poor tolerability in Part A of this study Part B may be conducted to explore higher doses using titration. Participants in both Parts A and B will participate in a 9 day wash-out period of current medication (Study Days 1-9); participants coming into the study on aripiprazole will remain on their current therapy throughout.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the safety and tolerability of escalating doses of LY2140023 in subjects with schizophrenia.

The secondary objectives of this study were:

* to characterize the pharmacokinetic (PK) parameters of LY2140023 and its active moiety - LY404039 in subjects with schizophrenia
* to explore higher doses of LY2140023 in subjects with schizophrenia for use in further regulatory studies
* to compare safety of LY2140023 to aripiprazole (ARP)
* to access changes in pharmacodynamic (PD) measures (Clinical Global Impression-Severity Scale [CGI-S], Extrapyramidal Symptoms [EPS], and Brief Psychiatric Rating Scale [BPRS])

This was an inpatient, open-label, multiple-dose, multi-center study to evaluate the safety and tolerability of LY2140023 given at doses expected to reflect multiples of the anticipated maximum therapeutic exposure under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of schizophrenic disorder
* Female participants who test negative for pregnancy at screening and agree to use a reliable method of birth control for the duration of the study and for at least 3 months after the last LY2140023 dose or are postmenopausal
* Not have been hospitalized for psychiatric illness for at least 12 weeks prior to Day 1 of washout period and have a Clinical Global Impression -Severity (CGI-S) scale score of <4
* Be willing and able as determined by the investigator to be hospitalized from the beginning of the washout period to the end of the study
* In the opinion of the investigator, the participant can be washed out of their Standard of Care (SOC) therapy (other than aripiprazole for the aripiprazole participants) for the duration of the study without detrimental effect to the participant's mental health (CGI-S <4 after completion of the washout period)
* Be considered reliable, have a level of understanding sufficient to perform all tests and examinations required by the protocol, and be willing to perform all study procedures
* Be able to understand the nature of the study and have given their own informed consent
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow blood sampling
* Clinically acceptable sitting blood pressure and pulse rate, as determined by the investigator

Participants on Aripiprazole prior to study entry must:

* On a stable dose of aripiprazole within the approved range in product labeling (less than or equal to 30 milligrams [mg]/day) for at least 60 days prior to Day 1 and with no anticipation of changes to dose, regimen (except as required for this study) or treatment within the next 1 month

Exclusion Criteria:

* Currently enrolled in, or discontinued within the 30 days prior to screening from, a clinical trial involving an investigational drug or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2140023, LY404039, aripiprazole, or related compounds
* Participants with moderate to severe renal impairment as defined by creatinine clearance (CrCl) <60 milliliters (mL)/minute (min)
* Have previously completed this study or have discontinued from any study investigating LY2140023 after having received at least 1 dose of LY2140023
* Participants for whom treatment with LY2140023 or aripiprazole as specified in this protocol, is relatively or absolutely clinically contraindicated
* Participants who have received treatment with clozapine
* Participants who have a diagnosis of schizophrenia who are taking either thioridazine or thiothixene
* Participants receiving treatment with depot antipsychotic medication within 12 weeks, prior to screening
* Participants who are taking any of medications that are specifically excluded
* Participants who have answered 'yes' to either Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the Columbia suicide severity rating scale (C-SSRS), or answer "yes" to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the "Suicidal Behavior" portion of the C-SSRS; and the ideation or behavior occurred within the past 3 months
* Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (Text Revision) (DSM-IV-TR) diagnosis of substance dependence or substance abuse (except nicotine and caffeine) within the 6 months prior to admission
* Diagnosis of substance-induced psychosis by DSM-IV-TR criteria within 7 days of admission (or at any time during the dosing period)
* Have a history of one or more seizures except for either of the following 2 situations: a single simple febrile seizure between ages 6 months and 5 years or a single seizure with an identifiable etiology, which has been completely resolved
* Have a screening electroencephalogram (EEG) with paroxysmal (epileptiform) activity, for example, one that demonstrates 3 or more focal sharp or spike waves, any sharp and slow wave complex, or any epileptiform discharge that is rhythmic, sustained, or generalized, or as locally defined
* Participants who have had electroconvulsive therapy (ECT) within 3 months of observation period or who are expected to have ECT at any time during the live phase of this study
* A diagnosis of Parkinson's disease, dementia-related psychosis, or related disorders
* Participant with untreated hyperthyroidism or hypothyroidism needing a thyroid hormone supplement who have not been on a stable dose of medication for at least 2 months prior to screening
* Have leukopenia or history of leukopenia during the participant's lifetime
* Participants with alanine aminotransferase (ALT/SGPT) or aspartate aminotransferase (AST/SGOT) values >2 times the upper limit of normal (ULN) of the performing laboratory, or total bilirubin values >1.5 times the ULN of the performing laboratory at screening
* Participants with corrected QT interval (Bazett's); QTcB >450 milliseconds (msec) (male) or >470 msec (female) at admission
* Have acute, serious or unstable medical conditions, including (but not limited to) inadequately controlled diabetes (hemoglobin A1c [HgbA1c] >8%), severe hypertriglyceridemia (fasting triglycerides greater than or equal to 500 milligrams/deciliter (mg/dL) or 5.65 micromoles/liter [umol/L]), hepatic insufficiency (specifically any degree of jaundice), recent cerebrovascular accidents, seizure disorders, serious acute systemic infection or immunology disease, unstable cardiovascular disorders (including ischemic heart disease), renal, gastroenterologic, respiratory, endocrinologic, neurologic, or hematologic diseases
* Prolactin level of >200 nanograms/milliliter (ng/mL) (200 micrograms/liter [ug/L], or 4228 milli international units/liter [mIU/L]) at screening with the exception of participants treated with risperidone. Participants treated with risperidone are excluded if the prolactin level is >300 ng/mL (300 ug/L, or 6342 mIU/L) at screening
* Participants with known medical history of Human Immunodeficiency Virus positive (HIV+) status
* Test positive for (1) Hepatitis C virus antibody or (2) Hepatitis B surface antigen (HBsAg) with or without positive Hepatitis B core total antibody. Participants with positive Hepatitis B core antibody test and negative HBsAg may be included in the study if ALT/SGPT and AST/SGOT levels are less than 2 times the ULN and total bilirubin does not exceed the ULN of the central laboratory

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-part study. The lead-in period was from Days 1 to 9, the test dosing (treatment) period was from Days 10 to 16, and the follow-up period was from Days 17 to 21. Dose escalation in Part A was completed. Part B (dose titration) was optional and not initiated because the objective of the study was met in Part A.
Groups:
- Aripiprazole: Participants continued current prescribed dosing regimen of orally administered aripiprazole (≤ 30 milligrams [mg]/day) from Study Day 1 to Study Day 21 (discharge).
- 160 mg LY2140023: 160 mg LY2140023 administered orally twice daily (BID) to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
- 240 mg LY2140023: 240 mg LY2140023 administered orally BID to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
- 320 mg LY2140023: 320 mg LY2140023 administered orally BID to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
- 400 mg LY2140023: 400 mg LY2140023 administered orally BID to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
- 480 mg LY2140023: 480 mg LY2140023 administered orally BID to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
Period: Overall Study
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Started | 16 | 12 (Included in this arm are six participants who erroneously received oral 80 mg LY2140023 BID.) | 11 | 12 | 12 | 12
Received at Least One Dose of Study Drug | 16 | 11 | 10 | 11 | 11 | 11
Completed | 13 | 11 | 9 | 7 | 11 | 6
Not Completed | 3 | 1 | 2 | 5 | 1 | 6
Not completed — Adverse Event | 1 | 0 | 0 | 4 | 0 | 5
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who were assigned to treatment and were either dosed or discontinued prior to dosing.
Groups:
- 160 mg LY2140023: 160 mg LY2140023 administered orally twice daily (BID) to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
  (Included in this arm are six participants who, rather than the assigned 160 mg BID LY2140023 dosage, erroneously received oral 80 mg LY2140023 BID on Study Days 10-15 and as a single, oral morning dose on Study Day 16.)
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023 | Total
Number analyzed (Participants) | 16 | 12 | 11 | 12 | 12 | 12 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (10) | 50 (7) | 49 (8) | 45 (10) | 42 (13) | 46 (10) | 45 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 2 | 2 | 1 | 3 | 18
  Male | 9 | 9 | 9 | 10 | 11 | 9 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 2 | 0 | 5
  Not Hispanic or Latino | 15 | 11 | 10 | 12 | 10 | 12 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 9 | 9 | 8 | 8 | 8 | 52
  White | 3 | 2 | 2 | 4 | 4 | 4 | 19
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 11 | 12 | 12 | 12 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Events (Physical Assessments and Clinical Lab Tests)
Description: Participants with at least 1 postdose (Day 10 through the end of study visit [Day 21]) treatment emergent adverse event (TEAE) were counted by dose cohort.
  A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to Day 21 for Part A
Population: Participants who were assigned to treatment and were either dosed or discontinued prior to dosing.
Measure: Number; unit: participants
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 16 | 12 | 11 | 12 | 12 | 12
participants
  Days 10-16 | 5 | 6 | 9 | 11 | 11 | 11
  Follow-up (Days 17-20) | 4 | 2 | 2 | 2 | 0 | 2
  End of Study (Day 21) | 1 | 1 | 1 | 1 | 0 | 1

2. Secondary Outcome: Part A: Pharmacokinetics, Maximum Concentration (Cmax)
Time Frame: Pre-dose and post-dose on Day 10 and Day 16
Population: Participants who received at least one dose of LY2140023 with evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- 160 mg LY2140023: 160 milligrams (mg) LY2140023 administered orally twice daily (BID) to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
  Not included in this arm are six participants who, rather than the assigned 160 mg BID LY2140023 dosage, erroneously received oral 80 mg LY2140023 BID on Study Days 10-15 and as a single, oral morning dose on Study Day 16.
Arm/Group | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 6 | 11 | 12 | 12 | 12
nanograms/milliliter (ng/mL)
  Day 10 (single dose): number analyzed (Participants) | 5 | 7 | 9 | 9 | 6
  Day 10 (single dose) | 496 (65) | 1170 (44) | 1410 (36) | 1830 (23) | 2630 (13)
  Day 16 (multiple doses): number analyzed (Participants) | 4 | 9 | 7 | 11 | 4
  Day 16 (multiple doses) | 799 (29) | 1090 (36) | 1510 (38) | 1760 (30) | 1810 (32)

3. Secondary Outcome: Part B: Pharmacokinetics, Maximum Concentration (Cmax)
Description: Part B (dose titration as defined in Part B of study) was not conducted because the objective of the study was met in part A.; therefore, no data are available for analysis of this secondary outcome
Time Frame: Pre-dose and post-dose on Days 12, 15, 18, 21, and 24
Population: Zero participants were analyzed.
Groups:
- 160 mg LY2140023: 160 milligrams (mg) LY2140023 administered orally twice daily (BID) to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
Arm/Group | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Part A: Pharmacokinetics, Area Under the Concentration - Time Curve (AUC)
Description: The Day 10 parameter is area under the concentration versus time curve from time zero to infinity (AUC[0-inf]) post-single dose of LY2140023. The Day 16 parameter is area under the concentration versus time curve in a dosing interval (AUC[0-tau]) post-repeated daily doses of LY2140023.
Time Frame: Pre-dose and post-dose on Day 10 and Day 16
Population: Participants who received at least one dose of LY2140023 with evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Groups:
- 160 mg LY2140023: 160 milligrams (mg) administered orally twice daily (BID) to participants on Study Days 10-15 and as a single, oral morning dose on Study Day 16. Administration of study drug included receiving the appropriate number of 80 mg LY2140023 tablets.
  Not included in this arm are six participants who, rather than the assigned 160 mg BID LY2140023 dosage, erroneously received oral 80 mg LY2140023 BID on Study Days 10-15 and as a single, oral morning dose on Study Day 16.
Arm/Group | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 6 | 11 | 12 | 12 | 12
nanograms*hours/milliliter (ng*hr/mL)
  Day 10 (single dose) (n=5, 7, 9, 9, 6): number analyzed (Participants) | 5 | 7 | 9 | 9 | 6
  Day 10 (single dose) (n=5, 7, 9, 9, 6) | 2800 (46) | 6290 (50) | 8100 (37) | 10600 (23) | 14700 (11)
  Day 16 (multiple doses) (n=4, 9, 7, 11, 4): number analyzed (Participants) | 4 | 9 | 7 | 11 | 4
  Day 16 (multiple doses) (n=4, 9, 7, 11, 4) | 4370 (21) | 6220 (32) | 7930 (39) | 9890 (28) | 10100 (31)

5. Secondary Outcome: Part B: Pharmacokinetics, Area Under the Concentration - Time Curve (AUC)
Description: Part B of this study was not conducted; therefore, no data are available for analysis.
Time Frame: Pre-dose and post-dose on Days 12, 15, 18, 21, and 24
Population: Zero participants were analyzed.
Arm/Group | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Increased Severity From Baseline to Day 17 in Clinical Global Impression- Severity Scale (CGI-S)
Description: Clinical Global Impression- Severity Scale (CGI-S) measures severity of illness at the time of assessment compared with start of treatment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The classification includes 1 = Normal, not at all ill, 2 = Borderline mentally ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, and 7 = Among the most extremely ill patients. Increases or higher scores indicate increasing severity (=worse outcome) Only incidences of selected shifts of increasing severity (an increase in numbers on a scale) were reported for participants.
  Part B of this study was not conducted; therefore, no data are available for analysis.
Time Frame: Baseline through Day 17 for Part A
Population: Participants who received at least one dose of LY2140023 with evaluable baseline and Day 17 Clinical Global Impression- Severity Scale data.
Measure: Number; unit: percentage of participants with shifts
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 16 | 11 | 10 | 11 | 11 | 11
percentage of participants with shifts
  Shift From Borderline to Mild | 0 | 0 | 0 | 9.1 | 0 | 0
  Shift from Mild to Moderate | 6.3 | 9.1 | 20.0 | 0 | 18.2 | 9.1

7. Secondary Outcome: Percentage of Participants With Worsening Symptoms From Baseline to Day 17 in Brief Psychiatric Rating Scale (BPRS)
Description: Brief Psychiatric Rating Scale (BPRS) is an 18-item clinician-administered scale used to assess the degree of severity of a participant's general psychopathological symptoms. Item scores ranged from 0 (not assessed) to 7 (extremely severe). Total Scores ranged from 0 to 126. Increases or higher scores indicate a worsening of symptoms.
  Only incidences of selected shifts of worsening symptoms (an increase in numbers on a scale within the 18-symptom construct) were reported for participants.
  Part B of this study was not conducted; therefore, no data are available for analysis.
Time Frame: Baseline through Day 17 for Part A
Population: Participants who received at least one dose of LY2140023 with evaluable baseline and Day 17 Brief Psychiatric Rating Scale data.
Measure: Number; unit: Percentage of participants with shifts
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 16 | 11 | 10 | 11 | 11 | 11
Percentage of participants with shifts
  Mild to moderately severe - Hallucinatory behavior | 12.5 | 0 | 0 | 0 | 0 | 0
  Mild to moderately severe - Anxiety | 0 | 0 | 10.0 | 0 | 0 | 0
  Very mild to moderate - Unusual thought content | 6.3 | 0 | 0 | 0 | 9.1 | 0
  Very mild to moderate - Excitement | 0 | 0 | 10.0 | 0 | 0 | 0
  Very mild to moderate - Conceptual disorganization | 0 | 0 | 0 | 0 | 9.1 | 0

8. Secondary Outcome: Percentage of Participants With Worsening Severity From Baseline to Day 17 in Extrapyramidal Symptoms as Measured by the Abnormal Involuntary Movement Scale (AIMS)
Description: The Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Increases or higher scores indicate a worsening of symptoms.
  The classification includes 0 = None, 1 = Minimal, may be extreme normal, 2 = Mild, 3 = Moderate, and 4 - Severe.
  Only incidences of selected shifts of worsening severity (an increase in numbers on a scale within the 10-item construct) were reported for participants.
  Part B of this study was not conducted; therefore, no data are available for analysis.
Time Frame: Baseline through Day 17 for Part A
Population: Participants who received at least one dose of LY2140023 with evaluable baseline and Day 17 Abnormal Involuntary Movement Scale data.
Measure: Number; unit: Percentage of participants with shifts
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 16 | 11 | 10 | 11 | 11 | 11
Percentage of participants with shifts
  Normal to Minimal - Jaw | 0 | 0 | 0 | 9.1 | 0 | 0
  Normal to Minimal - Muscles of facial expression | 0 | 0 | 0 | 0 | 9.1 | 0

9. Secondary Outcome: Percentage of Participants With Increasing Impairment From Baseline to Day 17 in Extrapyramidal Symptoms as Measured by the Simpson-Angus Scale (SAS)
Description: Simpson-Angus Scale (SAS) is used to measure Parkinsonian-type symptoms in participants exposed to antipsychotics. The scale consists of 10 items each rated on a 5-point scale, with 0 meaning complete absence of the condition and 4 meaning the presence of the condition in extreme form. The total score is obtained by adding the items. Increases or higher scores indicate a worsening of impairment.
  Only incidences of selected shifts of increasing impairment (an increase in numbers on a scale within the 10-symptom construct) were reported for participants.
  Part B of this study was not conducted; therefore, no data are available for analysis.
Time Frame: Baseline through Day 17 for Part A
Population: Participants who received at least one dose of LY2140023 with evaluable baseline and Day 17 Simpson-Angus Scale data.
Measure: Number; unit: Percentage of participants with shifts
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 16 | 11 | 10 | 11 | 11 | 11
Percentage of participants with shifts
  Normal to Slight - Gait | 6.3 | 0 | 0 | 0 | 0 | 0
  Normal to Slight - Head dropping | 6.3 | 0 | 0 | 0 | 0 | 0
  Normal to Slight - Tremor | 12.5 | 0 | 10.0 | 9.1 | 0 | 9.1
  Normal to Slight - Salivation | 6.3 | 0 | 0 | 0 | 0 | 0
  Normal to Slight - Glabella tap | 0 | 0 | 0 | 9.1 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Worsening Symptoms From Baseline to Day 17 in Extrapyramidal Symptoms as Measured by the Barnes Akathisia Scale (BAS)
Description: Barnes Akathisia Rating Scale (BAS) evaluates observable, restless movements of drug-induced akathisia associated with use of antipsychotic medications, includes objective (1-item) and subjective component (2-items, awareness of movement and distress related to movement) plus Global Clinical Assessment for overall disorder. Components were rated on a 4-point scale for the objective (0 = normal and 3 = constantly restless) and subjective items ((0 = absence of inner restlessness and 3 = awareness of intense compulsion to move for one item; and 0 = no distress and 3 = severe for the other item) and scored on a 6-point scale for the Global Clinical Assessment (0 = absent and 5 = severe). Increases or higher scores indicate a worsening of symptoms.
  Only incidences of selected shifts of worsening symptoms (an increase in numbers on a scale within the components) were reported for participants.
  Part B of this study was not conducted; therefore, no data are available for analysis.
Time Frame: Baseline through Day 17 for Part A
Population: Participants who received at least one dose of LY2140023 with evaluable baseline and Day 17 Barnes Akathisia Scale data.
Measure: Number; unit: Percentage of participants with shifts
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Number analyzed (Participants) | 16 | 11 | 10 | 11 | 11 | 11
Percentage of participants with shifts
  Objective - Normal to presence restless movements | 0 | 0 | 10.0 | 0 | 0 | 0
  Subjective - Awareness - Absence to non-specific | 0 | 0 | 10.0 | 9.1 | 9.1 | 9.1
  Subjective - Distress - No distress to mild | 0 | 0 | 10.0 | 0 | 0 | 0
  Global - Absent to questionable | 6.3 | 0 | 10.0 | 9.1 | 9.1 | 9.1

ADVERSE EVENTS:
Description: The analysis population included participants who received at least 1 dose of study drug (aripiprazole or LY2140023).
Arm/Group | Aripiprazole | 160 mg LY2140023 | 240 mg LY2140023 | 320 mg LY2140023 | 400 mg LY2140023 | 480 mg LY2140023
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/11 | 1/10 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 8/16 | 7/11 | 9/10 | 11/11 | 11/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Aripiprazole (N=16) | 160 mg LY2140023 (N=11) | 240 mg LY2140023 (N=10) | 320 mg LY2140023 (N=11) | 400 mg LY2140023 (N=11) | 480 mg LY2140023 (N=11)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 (0) | 0/9 (0) | 1/9 (1) | 0/10 (0) | 0 (0) | 0/9 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Aripiprazole (N=16) | 160 mg LY2140023 (N=11) | 240 mg LY2140023 (N=10) | 320 mg LY2140023 (N=11) | 400 mg LY2140023 (N=11) | 480 mg LY2140023 (N=11)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 8 (9) | 6 (9) | 4 (4) | 7 (13)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 6 (11) | 3 (8) | 9 (36)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electroencephalogram abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 5 (6) | 6 (10) | 6 (10) | 8 (8)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (4) | 2 (2) | 2 (2)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anticipatory anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/7 (0) | 0/3 (0) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 2/3 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (7) | 1 (1) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No analyses were performed and results were not calculated for Part B of this study because the study was stopped prior to Part B being initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days